CLINICAL TRIAL: NCT03360071
Title: A Double-blind, Prospective, Parallel Group Evaluation of a Novel Biologic Therapy for Perennial Allergic Rhinitis
Brief Title: A Novel Biologic Therapy for Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00107909
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Desensitization, Immunologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allergen Immunotherapy Group (Experimental)
  Interventions: Drug: Allergen Immunotherapy Extract
- Control Group (Placebo Comparator)
  Interventions: Drug: Allergen Immunotherapy Control

INTERVENTIONS:
Drug: Allergen Immunotherapy Extract — Allergen Immunotherapy treatment mixture to be delivered subcutaneously
  Arms: Allergen Immunotherapy Group
Drug: Allergen Immunotherapy Control — Allergen Immunotherapy Control Solution to be delivered subcutaneously
  Arms: Control Group

SUMMARY:
This is a randomized, parallel-group, double-blind, phase 2, single center, proof-of-concept study which will evaluate the effect of a preparation of FDA approved allergens (PMA) used as a sub-cutaneously administered immunotherapy for the management of allergic rhinitis (perennial and seasonal).

DETAILED DESCRIPTION:
This is a randomized, parallel-group, double-blind, phase 2, single center, proof-of-concept study which will evaluate the effect of a proprietory mixed preparation of FDA approved allergens (PMA) used as a sub-cutaneously administered immunotherapy for the management of allergic rhinitis (perennial and seasonal). Participating study subjects will be required to manifest the signs and symptoms of allergic rhinitis and test positive to at least six allergens using a multi aeroallergen screen at the time of study recruitment . All subjects will undergo standard allergen skin prick testing using six Multi-Test® PC skin prick test devices (Lincoln Diagnostics, Decator, IL) or comparable skin testing technique for a total of 48 Skin Prick Test (SPT). Approximately 36 total subjects will be enrolled.

Following a successful screening study visit and two week medication washout period, a 8 week treatment period will be initiated with bi-weekly study visits being undertaken, through to the end of immunotherapy, for assessment of therapeutic response and safety evaluations. Efficacy evaluation will be monitored using validated instruments that assess study subject clinical response, physician global assessment, and medication use. A safety assessment will be undertaken one month following completion of treatment.

At the screening visit (Screening Visit) a potential study subject will be required to fulfill the requirements of the study inclusion and exclusion criteria, will have a clinical evaluation including medical history and physical examination, blood draw and performance of skin testing. The study subject will then abstain from using intranasal steroids and antihistamines for two weeks and then return to the clinic for administration of sub-cutaneous PMA and post-treatment in-clinic safety evaluation. The latter evaluation period will comprise approximately 60 minutes to assess the study subject's response to PMA immunotherapy. Follow up clinic study visits will continue bi-weekly through 8 weeks and at each of these visits the study subject will receive increasing doses of PMA immunotherapy and will be evaluated for safety. Twice weekly clinical evaluation will also be performed. Following the final administration of PMA immunotherapy, a one month follow-up safety and clinical efficacy evaluation will be conducted by telephone or in the clinic. The duration of the study will be approximately 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements.
* The subject signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* The subject is a male or a non-pregnant, non-lactating female between the ages of 18 and 65.
* The subject is actively manifesting symptoms and signs of moderate to severe Perennial Allergic Rhinitis (PAR) with or without Seasonal Allergic Rhinitis (SAR) component defined as score of at least 28 on the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) and 6 on the Total Nasal Symptom Score (TNSS) scale. Scores will be determined on the first and second visit (after the 14 day medication washout period). Both scores exceeding their threshold on either day will qualify.
* Skin test strongly positive (wheal at least 5mm diameter and 2mm greater than negative control) to at least 6 of 48 allergy skin prick tests including at least one species of dust mite.

Exclusion Criteria:

* The subject has received any investigational compound within 30 days prior to screening.
* The subject has received allergen immunotherapy or Sublingual immunotherapy (SLIT) in a previous clinical study or as a therapeutic agent within the past two years.
* The subject has a history or clinical manifestations of significant medical conditions (cardiovascular, hepatic, infectious or renal disease, etc.) which in the opinion of the investigator renders them unacceptable study subjects.
* The subject has a history of drug abuse (defined as any chronic illicit drug use) or a history of alcohol abuse within 5 years prior to the screening visit.
* The subject is required to take excluded medications listed in Section 6.3.
* If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
* Subjects found to have on physical exam significant nasal polyps, septal deviation or infectious sinusitis.
* The subject has a history of allergic rhinitis but is not currently manifesting active signs and symptoms of the disorder.
* Subject has a history of cancer, other than squamous cell or basal cell carcinoma of the skin that has not been in full remission for at least 5 years prior to Screening. (A history of treated Cervical Intraepithelial Neoplasia (CIN) I, II, or CIN III is allowed.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allergen Immunotherapy Group | Control Group
Started | 17 | 14
Completed | 16 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergen Immunotherapy Group | Control Group | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (1) | 39 (1) | 36.8 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 8 | 6 | 14
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Daily Combined Score (DCS)
Description: Change in baseline. TNSS (Total Nasal Symptoms Score) + medication rescue score. TNSS is a scale of 0-12 with 12 being severe. Medication score is also 0-12 with 12 being highest use of medications. Thus DCS ranges from 0-24 (severe).
Time Frame: Change from baseline at 10 weeks
Measure: Mean (Standard Deviation); unit: DCS (daily combined score)
Arm/Group | Allergen Immunotherapy Group | Control Group
Number analyzed (Participants) | 17 | 14
DCS (daily combined score) | -4.41 (4.5) | -1.61 (3.2)

2. Primary Outcome: Mini RQLQ
Description: mini-RQLQ (mini-Rhinoconjunctivitis Quality of Life Questionnaire) is to measure a the level of severity of a set of symptoms of functional impairments due to rhinoconjunctivitis from baseline. 14 questions each range 0-6 (6 is most severe). Total range 0-84 (higher value is more severe symptoms).
Time Frame: Change from baseline at 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Allergen Immunotherapy Group | Control Group
Number analyzed (Participants) | 17 | 14
score on a scale | -34.9 (28.4) | -17.6 (9.8)

3. Secondary Outcome: Rescue Medication Use
Description: Use of epinephrine during intervention for a total of 8 weeks through followup and study completion (4 more weeks). Thus total number of times epinephrine is required per patient during entire 12 week period.
Time Frame: Duration of intervention plus followup (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Allergen Immunotherapy Group | Control Group
Number analyzed (Participants) | 17 | 14
Participants | 0 | 0

4. Secondary Outcome: Safety Assessment
Description: Safety and adverse events (AES) will be followed. We will measure and report systemic reactions.
Time Frame: continuous review of safety up to 14 week
Measure: Count of Participants; unit: Participants
Arm/Group | Allergen Immunotherapy Group | Control Group
Number analyzed (Participants) | 17 | 14
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: From start of therapy until one month after therapy was completed (12 weeks total).
Description: We look at all adverse events but particularly systemic reaction rates including anaphylaxis and use of epinephrine (12 weeks total)
Arm/Group | Allergen Immunotherapy Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 3/17 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allergen Immunotherapy Group (N=17) | Control Group (N=14)
systemic reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — mild systemic reaction defined by local inflammation and/or flushing or hives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication must be approved by sponsor within first 10 years after completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03360071/Prot_SAP_000.pdf